CLINICAL TRIAL: NCT04027985
Title: The Functional Outcome of Hemiplegic Upper Extremity in Patients With Subacute Stroke After Kinesiotaping Combined With Rehabilitation
Brief Title: Functional Outcome of Hemiplegic Upper Extremity in Patients With Subacute Stroke After Kinesiotaping and Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRPG8J0221
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-01

CONDITIONS: Stroke; Hemiplegia
Keywords: Kinesiotaping; Spasticity; Elastosonography; Stroke
MeSH Terms: conditions — Stroke; Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KT group (Experimental): the patients will receive KT for 5 days a week, for three weeks. And a 30-minute hand functional training would also be provided once daily every day during the intervention.
  Interventions: Other: Kinesiotaping; Other: Hand rehabilitation program
- Control group (Sham Comparator): the patients will receive sham KT for 5 days a week, for three weeks. And a 30-minute hand functional training would also be provided once daily every day during the intervention.
  Interventions: Other: Hand rehabilitation program; Other: Sham taping

INTERVENTIONS:
Other: Kinesiotaping — inesio tape would be applied over the extensor muscles of the affected hand for facilitating the extension of hand. We will apply the tape from the upper 1/3 length of dorsal side of the forearm and split the tape into five equal bars to the distal interphalangeal joint of each finger along the finger bones. This intervention would be executed for five days per week for three weeks.
  Arms: KT group
Other: Hand rehabilitation program — In the thirty-minute hand rehabilitation program, a motor-relearning theory would be implemented into the intervention by teaching the participants how to use their upper limb properly without any compensatory motions. Therefore, for establishing a correct movement pattern, an occupational therapist would provide a hand-guided activity, in which the participants could practice reaching movement as well as hand grasp and release in a more natural way. Besides, the therapist would also help the patients release their muscle tone by stretching the spastic muscles for five minutes before and after this hand rehabilitation period.
Other: Sham taping — A short piece of kinesio tape would be cut into half and applied over the lateral side of the forearm from the lateral epicondyle till the half of the forearm. The tape would not cover the both the flexor and extensor muscle bellies.
  Arms: Control group

SUMMARY:
1. To explore the role of sonoelastography with shear wave velocity to assess poststroke spasticity of affected arm and forearm muscles in patients with stroke.
2. To investigate the effects of Kinesiotaping applications on motor recovery, functional performance, and spasticity of affected upper extremity in patients with subacute stroke.

DETAILED DESCRIPTION:
Clinical characteristics of impaired motor performance on affected upper extremity in stroke patients included muscle weakness, increased muscle tone, contracture, joint instability, or impaired motor control. Poststroke spasticity (PSS) is also a common complication in stroke patients with limbs weakness and impaired coordination between agonist and antagonist contraction. Upper extremity impairments and PSS have negative effects on functional performances and quality of daily livings. In patients with subacute stroke, strengthening exercises, constraint-induce movement therapy, mirror therapy, mental practice, and neuromuscular electrical stimulation, botulinum toxin, and antidepressants are recommended. For managing PSS, several therapeutic interventions include stretching and range of motion exercises, antispasticity splint, neuromuscular electrical stimulation, oral medications, local injection with phenol or botulism, or surgery. Some investigators found that Kinesiotaping (KT) combined with other interventions may facilitate muscle function, provide joint support and proprioception feedback, and reduce pain in stroke patients with hemiplegia. The investigators will perform KT applications both on the proximal and distal parts of affected upper extremity to facilitate motor recovery and performance in subacute stroke patients with hemiplegia while receiving rehabilitation.

After reviewing literatures, sonoelastography and shear wave velocity (SWV) was applied to evaluate the muscle stiffness in stroke patients with upper limb spasticity, but mostly on biceps brachii muscle. The investigators try to use musculoskeletal sonography to explore the feasibility of sonoelastography as a quantitative tool for measuring PSS both on spastic arm and forearm muscles in patients with stroke.

In this study, sixty stroke patients with hemiplegia will be recruited for physical evaluations for PSS and functional performance of upper extremity, and sonoelastography with shear wave velocity (SWV) on biceps brachii, brachioradialis, flexor carpal radialis, and flexor carpal ulnaris muscles to explore the relationship between physical and sonographic assessements for PSS. In the next phase, 60 subacute patients with hemiplegia would be enrolled, then randomly divided into experimental or control groups. In experimental group (n=30), the patients will receive KT combined with rehabilitation once daily for five days, three weeks. In the control group (n=30), the patient will receive the same program without KT. All participants will receive following evaluations, including modified Ashworth and Tardieu scales, Fugl-Meyer Assessment for upper extremity, box and block test, the Wolf motor function test, and sonoelastography with shear wave velocity (SWV) before intervention, right after the three-week intervention, and three-week post intervention.

The aims of this study are:

1. To explore the role of sonoelastography with shear wave velocity to assess poststroke spasticity of affected arm and forearm muscles in patients with stroke.
2. To investigate the effects of Kinesiotaping applications on motor recovery, functional performance, and spasticity of affected upper extremity in patients with subacute stroke.

ELIGIBILITY:
Inclusion Criteria:

* The patients have a stroke with hemiplegia (duration is 3-6 months after stroke).
* Patients who are able to perform hand grasp.
* Patients who could slightly do fingers extension and minimal wrist extension. (ability of extension at least 10 degrees at the metacarpophalangeal and interphalangeal joints and 20 degrees at the wrist.)

Exclusion Criteria:

* age is younger than 18 years old or older than 80 years old;
* previous history of upper extremity tendon or neuromuscular injury;
* any other systemic neuromuscular disease; cognition or language impairment leading to communication difficulty.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
the change from baseline to time of MAS scale | 3rd week, and 6th week
  a therapist will measure spasticity of affected upper extremity at elbow and wrist joints (modified Ashworth scale). In this scale, muscle tone would be assessed by quick stretch of muscle belly. The scoring criteria are as follows. 0, no increase in muscle tone; 1, Slight increase in muscle tone; 2, More marked increase in muscle tone through most of the ROM; 3, considerable increase in muscle tone; 4, affected part(s) rigid in flexion or extension.
the change from baseline to time of Musculoskeletal sonography | 3rd week, and 6th week
  an experienced physiatrist will evaluate the findings on sonography, sonoelastography, and shear wave velocity (SWV). The participants will sit upright and put their upper extremities on the bed with elbow flexion in 90 degrees and the forearm full supination. The measured levels for evaluating FCR, FCU, and FDS muscles will be recorded at first time and use the same level at follow up for each patient. The SWV will be done in the longitudinal/transverse planes and be performed at the maximal cross-section area of the muscles and repeatedly measured for 7 times for each muscle. The sonoelastography will be applied in the longitudinal plane of the detected muscles at the same level of the SWV.
the change from baseline to time of Fugl-Meyer assessment for upper extremity | 3rd week, and 6th week
  a therapist will evaluate Fugl-Meyer assessment for upper extremity (FMA-UE) for each participant. In this assessment, participants would need to execute a series of movements, which involved proximal and distal part of upper limb. The higher the grade, the better the performance. The total score ranges from 0 to 66 for motor function.

SECONDARY OUTCOMES:
the change from baseline to time of Brunnstrom stage | 3rd week, and 6th week
  a therapist will measure motor recovery stage (Brunnstrom stage)
the change from baseline to time of modified Tardieu scale | 3rd week, and 6th week
  a therapist will measure spasticity of affected upper extremity at elbow and wrist joints (modified Tardieu scale).
the change from baseline to time of existence of sensation | 3rd week, and 6th week
  a therapist will measure the sensation, including light touch, pinprick touch, proprioception.
the change from baseline to time of quality of life by Stroke Impact Scale | 3rd week, and 6th week
  Stroke Impact Scale would be used to measure the independence of daily activities. It is a self-reported questionnaire. The contents involve various aspect of life. The high the grade, the more serious the life is affected. The total score is from 0 to 100 for self-assessing the level of recovery.
the change from baseline to time of quality of life by Barthel Index | 3rd week, and 6th week
  Barthel Index would be used to measure the independence of daily activities. It is a form that contains different activities of daily living. The higher the outcome grades, the better the level of independence.
the change from baseline to time of functional performance by box and block test | 3rd week, and 6th week
  box and block test would be used to assess the grasping and release performance of the affected hand.
the change from baseline to time of functional performance by STEF | 3rd week, and 6th week
  Simple Test for Evaluating Hand Function (STEF) would be used to assess the hand function by executing various types of grasping.

CONTACTS AND LOCATIONS:
Overall Officials: Yuchi Huang, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No